CLINICAL TRIAL: NCT04888195
Title: Symptom Clusters in Hong Kong Chinese Children With Blood Cancer:: A Longitudinal Study
Brief Title: Symptom Clusters in Hong Kong Chinese Children With Blood Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr Eva Ho, Assistant Professor, The Hong Kong Polytechnic University
Other Study IDs: SC_Blood_cancer
Record Dates: First submitted 2021-05-03; First posted 2021-05-17 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Child
Keywords: blood cancer; chemotherapy
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Questionnaire: This study aims to examine the cancer patient's symptom clusters and their changes over chemotherapy among pediatric patients with blood cancer in Hong Kong
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Participants will complete a set of validated questionnaires (TRSC-C and demographic sheet) before chemotherapy. They also have to complete the same questionnaires (TRSC-C) again within 1 week after the 1st, 2nd, 3rd, 4th , 5th and 6th courses of chemotherapy via telephone interview by our research assistants.

SUMMARY:
Pediatric blood cancer is the most common childhood malignancy. Despite its survival has been substantially improved, children still have to pay a high price for numerous distressing symptoms resulted from chemotherapy. Previous studies related to symptom experiences mainly focus on individual symptoms, rather than on multiple symptoms. Understanding these distressing symptoms may help healthcare professionals to develop appropriate and effective interventions with the aims of alleviating symptom severity and thus promoting the child's psychosocial well-being and quality of life.

DETAILED DESCRIPTION:
A longitudinal study design will be conducted. A sample of 120 patients age 5-17years, diagnosed with blood cancer but not yet receive any chemotherapy and able to communicate with Cantonese and read Chinese will be recruited in the pediatric oncology ward of Hong Kong Children's Hospital.

ELIGIBILITY:
Inclusion Criteria:

* aged 5 - 17 years old
* diagnosed with blood cancer but not yet receive any chemotherapy
* able to communicate with Cantonese and read Chinese

Exclusion Criteria:

* who are scheduled to have concurrent cancer treatment
* with recurrent malignancy
* medical condition, or cognitive and learning problems in their medical records

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: We will recruit pediatric patients with blood cancer in the Hong Kong Children's Hospital
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
The therapy-related symptom checklist for children (TRSC-C) | Before chemotherapy
  For measuring the occurrence and severity of symptoms experienced by patients aged 5-17 when they undergo cancer treatment.
The therapy-related symptom checklist for children (TRSC-C) at 1-week | At 1-week follow-up
  For measuring the occurrence and severity of symptoms experienced by patients aged 5-17 when they undergo cancer treatment.
The therapy-related symptom checklist for children (TRSC-C) at 1-month | At 1-month follow-up
  For measuring the occurrence and severity of symptoms experienced by patients aged 5-17 when they undergo cancer treatment.
The therapy-related symptom checklist for children (TRSC-C) at 3-month | At 3-month follow-up
  For measuring the occurrence and severity of symptoms experienced by patients aged 5-17 when they undergo cancer treatment.
The therapy-related symptom checklist for children (TRSC-C) at 6-month | At 6-month follow-up
  For measuring the occurrence and severity of symptoms experienced by patients aged 5-17 when they undergo cancer treatment.
Demographic sheet | At baseline
  collect the background information of our subjects, including their age, gender, educational attainment, parents' marital status and religious belief

CONTACTS AND LOCATIONS:
Overall Officials: Ka Yan Ho, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- Ka Yan Ho, Hong Kong, Hong Kong,China, Hong Kong

IPD SHARING:
Plan to Share IPD: No